CLINICAL TRIAL: NCT04525313
Title: The Prediction Model of Avastin Plus Chemotherapy as First Line Treatment in Unresectable Ras Mutant Colorectal Liver Metastase (CRLM) Patients
Brief Title: The Prediction Model of Avastin Plus Chemotherapy in Unresectable Ras Mutant CRLM Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: BECOME1
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — primary tumor proteins of CRLM patients before avastin plus chemotherapy treatment will be sequenced by mass spectrum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training set: 58 unresectable simutaneous CRLM patients with ras mutation accepted Avastin plus chemotherapy treatment after primary tumor resection between 2013.01 and 2017.12.
- validation set: another 58 unresectable simutaneous CRLM patients with ras mutation accepted Avastin plus chemotherapy treatment after primary tumor resection between 2018.01 and 2022.12.

SUMMARY:
establishment and validation of the prediction model of avastin plus chemotherapy as first line treatment in simultaneous ras mutant unresectable CRLM patients

DETAILED DESCRIPTION:
Ras mutant unresectable CRLM patients with primary tumor resection followed by avastin in combination with chemotherapy were included in this study. The tumor response was assessed by local MDT group. Based on tumor response, 58 CRLM patients were classified into two groups (CR+PR vs SD+PD). Primary samples of the two group patients will be sequenced by mass spectrum. After MS sequencing, a prediction model will be estimated. Another 58 CRLM patients will be inclued for validation of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

age 18-75 years, histologically proven colorectal adenocarcinoma, with liver-dominant disease, a life expectancy of > 3 months, ras mutation, unresectable simultaneous liver metastasis, ECOG 0-1, written informed consent for participation in the trial.

Exclusion Criteria:

patients with known hypersensitivity reactions to any of the components of the study treatments, pregnancy or breast-feeding, accepted chemotherapy, radiotherapy and target therapy before primary tumor resection, other previous malignancy within 5 years, known drug abuse/alcohol abuse, ECOG>1, legal incapacity or limited legal capacity.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Simultaneous unresectable CRLM patients(ras mutation) with primary tumor resection before Avastin plus chemotherapy as first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
response rate | 6 months
  response rate will be assessed by local MDT every two months

SECONDARY OUTCOMES:
overall survival | 3 years
  overall survival will be assessed by researchers every two months during treatment, and telephone follow-up every three month after treatment
progression free survival | 3 years
  progression free survival will be assessed by local MDT every two months during treatment, and telephone follow-up every three month after treatment

IPD SHARING:
Plan to Share IPD: Undecided